CLINICAL TRIAL: NCT07041996
Title: Mobile Phone-Based Sarcopenia Screening Application for Early Detection of Sarcopenia
Brief Title: Sarcopenia Screening Application for Sarcopenia
Status: Not yet recruiting | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Irma Ruslina Defi, Principal Investigator, Universitas Padjadjaran
Other Study IDs: IKFR.12.06.25
Record Dates: First submitted 2025-06-13; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Geriatrics Rehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults (≥60 years) visiting the Geriatric Clinic: Patients aged over 60 years completed the SARC-F questionnaire in the mobile application to assess the risk of sarcopenia
  Interventions: Diagnostic Test: Mobile-based SARC-F screening application

INTERVENTIONS:
Diagnostic Test: Mobile-based SARC-F screening application — SARC-F mobile application as a digital health intervention for sarcopenia risk assessment.

SUMMARY:
Patients aged over 60 years completed the SARC-F questionnaire in the mobile application to assess the risk of sarcopenia.

DETAILED DESCRIPTION:
Patients aged over 60 years completed the SARC-F questionnaire in the mobile application to assess the risk of sarcopenia. The aim of this study was to develop a mobile application for self-screening of sarcopenia in the elderly specifically in Indonesia using the SARC-F questionnaire. This application is expected to improve accessibility, cost-effectiveness, and ease of health education, enabling early detection and rapid intervention to reduce the disease burden of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in this study
* Patients over 60 years old with or without caregivers
* Patients with or without caregivers with a mobile phone
* Agree to participate in the black-box testing and sign the informed consent form
* Complete the whole sequence of the trial

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The accessible population is patients over 60 years of age who visit Geriatric Polyclinic in Bandung
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia status in mobile phone applications | 6 month
  Using Sarcopenia Questionnaire (SARC-F), score in numerical 0-10